CLINICAL TRIAL: NCT00229255
Title: Relation of Obesity With Frequency of Meals (MST 0557)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MST-0557
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Obesity; Insulin Resistance; Fatty Liver
Keywords: Non-Alcoholic hepatic steatosis
MeSH Terms: conditions — Obesity; Insulin Resistance; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high frequency meals group (Active Comparator): High carbohydrate diet i.e. 65% carbohydrate, 15% protein, 20% fat for 4 weeks.
  Interventions: Other: high frequency of meals
- twice-a -day meals (Active Comparator): high carbohydrate diet i.e. 65% carbohydrate, 15% protein, 20% fat for 4 weeks
  Interventions: Other: twice a day meals

INTERVENTIONS:
Other: high frequency of meals — high carbohydrate diet i.e. 65% carbohydrate, 15% protein, 20% fat for 4 weeks.
  Arms: high frequency meals group
Other: twice a day meals — high carbohydrate diet i.e. 65% carbohydrate, 15% protein, 20% fat for 4 weeks.
  Arms: twice-a -day meals

SUMMARY:
The purpose of this study is to test the relationship between frequency of meals and hepatic fat content and insulin sensitivity. We, the researchers at Rockefeller University, hypothesize that low plasma insulin levels (as achieved by periods of fasting) will prevent insulin resistance and reduce hepatic lipid content. In contrast, frequent, carbohydrate-rich meals will predispose to hepatic steatosis (non-alcoholic) and insulin resistance.

This is a 6 week inpatient study.

DETAILED DESCRIPTION:
The hypothesis will be tested by studying two groups of normal subjects who will receive a defined weight maintenance diet: one group will be given meals twice a day and other group will be given eight meals (snacks) per day. At the beginning of the study period and after 4 weeks following the specified frequency of meals, the study subjects will have their whole body insulin sensitivity and hepatic fat content measured by the euglycemic-hyperinsulinemic clamp and MRI of the liver, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals
2. Age between 18-45 years
3. Body mass index (BMI) between 18.5 - 24.9

Exclusion Criteria:

1. Diabetes mellitus
2. Chronic drug treatment for any medical condition like hypertension or hyperlipidemia, hyperthyroidism or taking weight control medications.
3. Inability to give informed consent.
4. Inability to give contact information including permanent residence or provide evidence of stable living environment for the study period.
5. Active weight reduction of more than 7 pounds in the last 3 months.
6. History of bleeding or blood clotting disorders.
7. Pregnancy or breast-feeding in the women.
8. History of anaphylaxis or anaphylactoid-like reaction as a result of food allergies.
9. HIV or hepatitis B and C positive subjects.
10. Subjects with hemoglobin < 8.5 gm/dl.
11. Abnormal liver function test (ALT, AST, alkaline phosphate, LDH, GGT or total bilirubin).
12. Serum creatinine or BUN greater than the upper limit of the normal, serum albumin less than 3.5g/dl, or proteinuria 1+ or greater.
13. History of alcohol intake of more than 40 g/day.
14. Contraindications to magnetic resonance imaging (MRI) including pacemakers, surgical clips, metallic implants, neuromuscular- skeletal stimulators and internal orthopedic screws or rods.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2005-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
We will determine total body insulin sensitivity with the help of the hyperinsulinemic-euglycemic clamp. We will also assess hepatic steatosis by conducting MRI scans on our subjects. | days 8,9,11 41 and 42

SECONDARY OUTCOMES:
Weight, waist and hip circumference, fasting glucose and insulin, serum ketones, lipids and lipoproteins including VLDL and apolipoprotien B100, liver function tests, serum adiponectin (marker for insulin resistance), and measures of hunger. | days 1-42

CONTACTS AND LOCATIONS:
Overall Officials: Markus Stoffel, MD, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States